CLINICAL TRIAL: NCT02643693
Title: User Acceptability of a Nicotine Lactate Delivery System Relative to the VUSE e-Cigarette System and Combustible Cigarette Comparators
Brief Title: User Acceptability of a Nicotine Lactate Delivery System (P3L)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P3L-PK-02-US
Record Dates: First submitted 2015-12-17; First posted 2015-12-31 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Smoking
Keywords: Conventional cigarette; Nicotine lactate delivery system; e-cigarette; VUSE; Combustible cigarette
MeSH Terms: conditions — Smoking; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- P3L Product use (Experimental): Subject product use was randomly assigned for each ad libitum use session, following a sequence of product exposure comprised of the three products (P3L, VUSE, and CC).
  Interventions: Other: P3L
- VUSE Product Use (Experimental): Subject product use was randomly assigned for each ad libitum use session, following a sequence of product exposure comprised of the three products (P3L, VUSE, and CC).
  Interventions: Other: VUSE
- CC Product Use (Experimental): Subject product use was randomly assigned for each ad libitum use session, following a sequence of product exposure comprised of the three products (P3L, VUSE, and CC).
  Interventions: Other: CC

INTERVENTIONS:
Other: P3L — Ad libitum use for a maximum of three hours.
  P3L delivers, on average, 80 µg of nicotine per puff under Health Canada Intense smoking regime.
  Arms: P3L Product use
Other: VUSE — Ad libitum use for a maximum of three hours.
  VUSE delivers, on average, 80 µg of nicotine per puff based on the CORESTA e-cigarette recommended smoking regime.
  Arms: VUSE Product Use
Other: CC — Ad libitum use of the subject's own brand of non-menthol CC for a maximum of three hours.
  Arms: CC Product Use

SUMMARY:
This study will provide an initial assessment of the acceptability of the Nicotine Lactate Delivery System (P3L) after ad libitum use and the ability of combustible cigarette (CC) smokers to use P3L to maintain their customary nicotine intake, in a manner comparable with their own brand of CC or the VUSE e-cigarette system.

DETAILED DESCRIPTION:
The total duration of the study for an individual subject will be between 3 and 8 weeks, including 1 day for the screening visit, 3 days for the ad libitum use sessions (P3L, VUSE e-cigarette system and subjects' own commercially available non-menthol CC), 1 day for the preference evaluation session (subjects will be given the choice of using ad libitum the P3L or the VUSE), the 2 to 10 days of interval between each visit, and 7 days for the passive safety follow-up period.

The pharmacokinetics (PK) and pharmacodynamics (PD, i.e., subjective effects) profiles, will be evaluated as well as the safety and tolerability of the P3L.

ELIGIBILITY:
Inclusion Criteria:

* Smoking, healthy subject as judged by the Investigator
* Subject smoked at least 10 commercially available non-menthol CCs per day for the last 12 months
* Subject does not plan to quit smoking in the next 60 days

Exclusion Criteria:

* As per Investigator judgment, the subject cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason)
* Subject has donated or been in receipt of whole blood or blood products within 3 months prior to the screening visit
* Subject has used tobacco products or nicotine containing products other than CCs within 30 days prior to the screening visit
* Female subject is pregnant or breast feeding
* Female subject does not agree to use an acceptable method of effective contraception
* Female subject uses estrogen-containing hormonal contraception or hormone replacement therapy

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.; Jed E. Rose, PhD, Principal Investigator — Rose Research Center, LLC
Locations (1):
- Rose Research Center, LLC, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox LS, Tiffany ST, Christen AG. Evaluation of the brief questionnaire of smoking urges (QSU-brief) in laboratory and clinical settings. Nicotine Tob Res. 2001 Feb;3(1):7-16. doi: 10.1080/14622200020032051. PMID 11260806

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated (1st subject screened): 16 November 2015 A demonstration of the P3L system and the VUSE e-cigarette system was given to the subjects.
Pre-assignment Details: Enrolled population = 24 subjects All enrolled subjects met all of the inclusion and none of the exclusion criteria for the study.
  Subject product use was randomly assigned for each ad libitum use session, following a sequence of product exposure comprised of the three products (P3L, VUSE, and CC).
Groups:
- P3L/Vuse/CC Product Exposure: Subjects followed a sequence of product exposure comprised of P3L; VUSE; CC.
- P3L/CC/Vuse Product Exposure: Subjects followed a sequence of product exposure comprised of P3L; CC; Vuse.
- Vuse/CC/P3L Product Exposure: Subjects followed a sequence of product exposure comprised of Vuse; CC; P3L.
- Vuse/P3L/CC Product Exposure: Subjects followed a sequence of product exposure comprised of Vuse; P3L; CC.
- CC/P3L/Vuse Product Exposure: Subjects followed a sequence of product exposure comprised of CC; P3L; Vuse.
- CC/Vuse/P3L Product Exposure: Subjects followed a sequence of product exposure comprised of the three products (CC; Vuse; P3L).
Period: Overall Study
Arm/Group | P3L/Vuse/CC Product Exposure | P3L/CC/Vuse Product Exposure | Vuse/CC/P3L Product Exposure | Vuse/P3L/CC Product Exposure | CC/P3L/Vuse Product Exposure | CC/Vuse/P3L Product Exposure
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 2 | 2 | 3 | 4 | 4 | 3
Not Completed | 2 | 2 | 1 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Adherence Issues | 2 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects who gave informed consent and had exposure to at least one of the investigational products as part of the study (including P3L system, the VUSE e-cigarette system or CC).
Groups:
- P3L/VUSE/CC Product Exposure: Subject product use was randomly assigned for each ad libitum use session, following a sequence of product exposure comprised of the three products (P3L, VUSE, and CC).
Arm/Group | P3L/VUSE/CC Product Exposure
Number analyzed (Participants) | 22
Age, Customized [Count of Participants; unit: Participants]
  <=19 years | 0
  Between 19 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Plasma Concentration of Nicotine/Cotinine After Each ad Libitum Use Session.
Description: For each ad libitum use session (P3L, VUSE, and CC), change from baseline plasma concentration of Nicotine/Cotinine was measured from two blood samples collected before product use (to provide baseline measures) and from two blood samples collected following product use (to show change from baseline).
Time Frame: Measured at 15 minutes and 5 minutes prior to each 3 hour product use to provide baseline measures, then at 15 minutes and 30 minutes after product use period to show change from baseline.
Population: All the subjects who gave informed consent and completed all three ad libitum use sessions, without major protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: (ng/mL)
Groups:
- P3L Product Exposure; VUSE Product Exposure; CC Product Exposure: Subject product use was randomly assigned for each ad libitum use session, following a sequence of product exposure comprised of the three products (P3L, VUSE, and CC).
Arm/Group | P3L Product Exposure | VUSE Product Exposure | CC Product Exposure
Number analyzed (Participants) | 16 | 16 | 16
(ng/mL)
  Baseline (Average) before session: Nicotine | 1.7621 [1.1308 to 2.7459] | 2.4113 [1.8529 to 3.1378] | 1.9446 [1.5375 to 2.4594]
  Change from Baseline after session: Nicotine | 5.5571 [3.5802 to 8.6255] | 7.3425 [4.7138 to 11.4371] | 17.1821 [13.7633 to 21.4500]
  Baseline (Average) before session: Cotinine | 182.554 [148.073 to 225.065] | 187.559 [147.914 to 237.828] | 199.547 [161.636 to 246.351]
  Change from Baseline after session: Cotinine | 15.222 [10.116 to 22.905] | 11.163 [5.523 to 22.561] | 33.888 [24.004 to 47.842]

2. Primary Outcome: Overall Score of the Short Version of the Questionnaire of Smoking Urges (QSU-brief). Total Score; Factor 1 (Reward); Factor 2 (Relief)
Description: The QSU-Brief questionnaire is an instrument used to measure urge to smoke. Subjects were asked to respond to 10 questions, scored from 1 to 7 on a 7-point scale. A score of 1 on this scale indicates a very low urge to smoke, while a score of 7 indicates a very high urge to smoke. Subjects were asked to complete the questionnaire before, during, and after each ad libitum product use session. (P3L, VUSE, and Subjects' Own Brand of Non-menthol CC).
  Two factor scores and a total score were derived. Factor 1 represents the desire and intention to smoke with smoking perceived as rewarding, while Factor 2 represents an anticipation of relief from negative effect with an urgent desire to smoke.
  Products were compared over all timepoints using a repeated measure model using values after t0.
  The model adjusted for baseline value, sequence, and period with repeated measure over time and a random effect in subjects. Adjusted mean over all timepoints, for each timepoint, were estimated.
Time Frame: QSU-brief questionnaire completed before product use session, then at 60 mins, 120 mins, and 180 mins after starting each product use session.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | P3L Product Exposure | VUSE Product Exposure | CC Product Exposure
Number analyzed (Participants) | 16 | 16 | 16
score on a scale
  Total Score - Over all timepoints | 3.86 [3.36 to 4.36] | 3.08 [2.58 to 3.58] | 1.93 [1.43 to 2.42]
  Total Score - t0 + 60mins | 4.02 [3.51 to 4.52] | 3.24 [2.74 to 3.74] | 2.09 [1.58 to 2.59]
  Total Score - t0 + 120mins | 3.84 [3.33 to 4.36] | 3.07 [2.56 to 3.58] | 1.91 [1.40 to 2.42]
  Total Score - t0 + 180mins | 3.71 [3.20 to 4.23] | 2.94 [2.42 to 3.45] | 1.78 [1.27 to 2.29]
  Factor 1 - Over all timepoints | 4.97 [4.39 to 5.54] | 4.11 [3.54 to 4.68] | 2.15 [1.58 to 2.73]
  Factor 1 - t0 + 60mins | 4.87 [4.28 to 5.46] | 4.48 [3.89 to 5.06] | 2.53 [1.94 to 3.12]
  Factor 1 - t0 + 120mins | 4.99 [4.33 to 5.64] | 4.11 [3.46 to 4.77] | 2.08 [1.42 to 2.74]
  Factor 1 - t0 + 180mins | 5.05 [4.43 to 5.66] | 3.74 [3.13 to 4.35] | 1.84 [1.23 to 2.46]
  Factor 2 - Over all timepoints | 2.85 [2.34 to 3.36] | 2.15 [1.64 to 2.66] | 1.60 [1.10 to 2.11]
  Factor 2 - t0 + 60mins | 2.95 [2.43 to 3.48] | 2.25 [1.73 to 2.78] | 1.71 [1.19 to 2.23]
  Factor 2 - t0 + 120mins | 2.84 [2.33 to 3.35] | 2.14 [1.63 to 2.65] | 1.59 [1.09 to 2.10]
  Factor 2 - t0 + 180mins | 2.76 [2.24 to 3.28] | 2.06 [1.54 to 2.58] | 1.51 [1.00 to 2.03]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the entire study duration of up to 5 months, with individual subject participation of between three and 11 weeks from the signature of the Informed Consent Form (ICF) until the end of the safety follow-up period.
Description: The safety was assessed in the safety population, consisting of all randomized subjects who gave informed consent and had exposure to at least one of the investigational products as part of the study (including P3L system, the VUSE e-cigarette system or CC).
  Overall safety population = 22 subjects; P3L exposure = 21 subjects; VUSE exposure = 19 subjects; CC exposure = 19 subjects.
Groups:
- P3L Product; VUSE Product; CC Product: Subject product use was randomly assigned for each ad libitum use session, following a sequence of product exposure comprised of the three products (P3L, VUSE, and CC).
Arm/Group | P3L Product | VUSE Product | CC Product
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 14/21 | 13/19 | 9/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P3L Product (N=21) | VUSE Product (N=19) | CC Product (N=19)
Headache (Nervous system disorders) | 4 (4) | 3 (3) | 2 (2)
Disturbance In Attention (Nervous system disorders) | 3 (4) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 6 (8) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 1 (1)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0)
Feeling Jittery (General disorders) | 5 (5) | 4 (4) | 2 (2)
Chest Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Unevaluable Event (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.